CLINICAL TRIAL: NCT05566288
Title: A Four Way Crossover Thorough QT/QTc Study to Evaluate the Electrocardiographic Effects of Therapeutic and Supratherapeutic Doses of Cytisinicline in Healthy Smokers
Brief Title: Study to Evaluate Electrocardiographic Effects of Therapeutic & Supratherapeutic Doses of Cytisinicline in Healthy Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ACH-CYT-06
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the moxifloxacin treatment will not be blinded to site personnel and the participants, but moxifloxacin treatment will be blinded to the central cardiologist for assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Sequence 1 (Experimental): Participants will receive the assigned study drug after an overnight fast on Day 1 during each of 4 periods in the following order:
  * Cytisinicline, 6 mg (therapeutic dose) (2 cytisinicline tablets+6 placebo tablets)
  * Cytisinicline, 24 mg (supratherapeutic dose) (8 cytisinicline tablets)
  * Placebo (negative control) (8 placebo tablets)
  * Moxifloxacin 400 mg PO (positive control) (1 tablet) There will be a minimum 5 day washout between dosing periods.
  Interventions: Drug: Cytisinicline; Drug: Placebo; Drug: Moxifloxacin
- Sequence 2 (Experimental): Participants will receive the assigned study drug after an overnight fast on Day 1 during each of 4 periods in the following order:
  * Cytisinicline, 24 mg (supratherapeutic dose) (8 cytisinicline tablets)
  * Moxifloxacin 400 mg PO (positive control) (1 tablet)
  * Cytisinicline, 6 mg (therapeutic dose) (2 cytisinicline tablets+6 placebo tablets)
  * Placebo (negative control) (8 placebo tablets) There will be a minimum 5 day washout between dosing periods.
  Interventions: Drug: Cytisinicline; Drug: Placebo; Drug: Moxifloxacin
- Sequence 3 (Experimental): Participants will receive the assigned study drug after an overnight fast on Day 1 during each of 4 periods in the following order:
  * Placebo (negative control) (8 placebo tablets)
  * Cytisinicline, 6 mg (therapeutic dose) (2 cytisinicline tablets+6 placebo tablets)
  * Moxifloxacin 400 mg PO (positive control) (1 tablet)
  * Cytisinicline, 24 mg (supratherapeutic dose) (8 cytisinicline tablets) There will be a minimum 5 day washout between dosing periods.
  Interventions: Drug: Cytisinicline; Drug: Placebo; Drug: Moxifloxacin
- Sequence 4 (Experimental): Participants will receive the assigned study drug after an overnight fast on Day 1 during each of 4 periods in the following order:
  * Moxifloxacin 400 mg PO (positive control) (1 tablet)
  * Placebo (negative control) (8 placebo tablets)
  * Cytisinicline, 24 mg (supratherapeutic dose) (8 cytisinicline tablets)
  * Cytisinicline, 6 mg (therapeutic dose) (2 cytisinicline tablets+6 placebo tablets) There will be a minimum 5 day washout between dosing periods.
  Interventions: Drug: Cytisinicline; Drug: Placebo; Drug: Moxifloxacin
- Sequence 5 (Experimental): Participants will receive the assigned study drug after an overnight fast on Day 1 during each of 4 periods in the following order:
  * Cytisinicline, 24 mg (supratherapeutic dose) (8 cytisinicline tablets)
  * Placebo (negative control) (8 placebo tablets)
  * Cytisinicline, 6 mg (therapeutic dose) (2 cytisinicline tablets+6 placebo tablets)
  * Moxifloxacin 400 mg PO (positive control) (1 tablet) There will be a minimum 5 day washout between dosing periods.
  Interventions: Drug: Cytisinicline; Drug: Placebo; Drug: Moxifloxacin
- Sequence 6 (Experimental): Participants will receive the assigned study drug after an overnight fast on Day 1 during each of 4 periods in the following order:
  * Placebo (negative control) (8 placebo tablets)
  * Moxifloxacin 400 mg PO (positive control) (1 tablet)
  * Cytisinicline, 24 mg (supratherapeutic dose) (8 cytisinicline tablets)
  * Cytisinicline, 6 mg (therapeutic dose) (2 cytisinicline tablets+6 placebo tablets) There will be a minimum 5 day washout between dosing periods.
  Interventions: Drug: Cytisinicline; Drug: Placebo; Drug: Moxifloxacin
- Sequence 7 (Experimental): Participants will receive the assigned study drug after an overnight fast on Day 1 during each of 4 periods in the following order:
  * Cytisinicline, 6 mg (therapeutic dose) (2 cytisinicline tablets+6 placebo tablets)
  * Cytisinicline, 24 mg (supratherapeutic dose) (8 cytisinicline tablets)
  * Moxifloxacin 400 mg PO (positive control) (1 tablet)
  * Placebo (negative control) (8 placebo tablets) There will be a minimum 5 day washout between dosing periods.
  Interventions: Drug: Cytisinicline; Drug: Placebo; Drug: Moxifloxacin
- Sequence 8 (Experimental): Participants will receive the assigned study drug after an overnight fast on Day 1 during each of 4 periods in the following order:
  * Moxifloxacin 400 mg PO (positive control) (1 tablet)
  * Cytisinicline, 6 mg (therapeutic dose) (2 cytisinicline tablets+6 placebo tablets)
  * Placebo (negative control) (8 placebo tablets)
  * Cytisinicline, 24 mg (supratherapeutic dose) (8 cytisinicline tablets) There will be a minimum 5 day washout between dosing periods.
  Interventions: Drug: Cytisinicline; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Cytisinicline — compressed film-coated tablet containing 3 mg cytisinicline
  Other Names: Cytisine
Drug: Placebo — Placebo tablets to match compressed film-coated tablet containing 3 mg cytisinicline
Drug: Moxifloxacin — 400 mg tablets

SUMMARY:
The primary objective of this trial is to assess the effects of cytisinicline at therapeutic and supratherapeutic doses on cardiac repolarization relative to placebo in healthy adult subjects who are smokers.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the following criteria to be eligible for inclusion into the study:

1. Regular moderate cigarette smokers (minimum 10 cigarettes per day).
2. Healthy males and females 18-45 years of age.
3. If woman, she meets one of the following criteria:

   1. is of non-childbearing potential (refer to Section 8.3-Contraception Requirements for the criteria for non-childbearing potential status); or
   2. is of childbearing potential and agrees to use an accepted contraceptive method (refer to Section 8.3-Contraception Requirements for a list of accepted methods) from at least 4 weeks prior to admission to period 1 until at least the last study drug administration.
4. No clinically significant abnormal serum chemistry or hematology values at Screening.
5. Body mass index (BMI) within 18-30 kg/m2 at Screening.
6. Subject must be willing to communicate with the investigator and site staff and comply with all study procedures and requirements.
7. Subject must be able to provide written, informed consent including compliance with the requirements listed in the consent form.
8. Subject must be able and willing to swallow whole tablets without breaking, cutting, or chewing.

Exclusion Criteria:

Subjects meeting ANY of the following exclusion criteria will NOT be eligible for inclusion into the study.

1. History or presence of a systemic disease, which as judged by the investigator, may affect the subject's ability to participate in the study or in the outcome of the study.
2. Evidence of infection with Hepatitis B or C, or human immunodeficiency virus HIV-1 or HIV-2, as determined by results of testing at Screening.
3. Female subjects who are pregnant or lactating.
4. Family history of QTc prolongation or of unexplainable sudden death at <50 years of age.
5. History of QTc prolongation or knowledge of any kind of cardiovascular disorder/condition known to increase the possibility of QT prolongation or history of additional risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome or Brugada Syndrome) or cardiac conduction disorders.
6. History of myocardial infarction, unstable angina pectoris, cerebrovascular disease, atherosclerosis or arterial hypertension.
7. History of rare hereditary problem of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
8. History of glucose 6-phosphate dehydrogenase deficiency or myasthenia gravis.
9. Use of any medication that might interfere with the PK of cytisinicline.
10. Resting supine pulse rate less than 50 beats per minute or greater than 100 beats per minute at Screening.
11. Resting supine systolic blood pressure less than 90 mmHg or greater than 140 mmHg; resting supine diastolic blood pressure less than 50 mmHg or greater than 90 mmHg at Screening.
12. Clinically significant ECG abnormalities at Screening, including:

    1. QTcF >450 ms
    2. QRS >110 ms
    3. PR >200 ms
    4. Second or third-degree atrioventricular (AV) block
    5. Any rhythm other than sinus rhythm, which is interpreted by the investigator to be clinically significant
13. Renal impairment defined as a creatinine clearance (CrCl) <90 mL/min, based on creatinine clearance calculation by the Cockcroft-Gault formula and normalized to an average surface area of 1.73 m2, at Screening.
14. Serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) above the ULN (upper limit of the reference range at Screening).
15. Positive urine drug and alcohol screen at Screening or Day -1 for each Treatment Period.
16. Positive pregnancy test for women of child-bearing potential (WOCBP) at Screening or Day-1 to each Treatment Period.
17. History of significant alcohol abuse, drug abuse, or use of illicit drugs within one year prior to Screening.
18. Average weekly alcohol consumption of >14 units for males and >7 units for females within the previous 6 months.
19. Average daily consumption of methylxanthines-containing beverages or food (e.g., coffee, tea, cola, sodas, chocolate) equivalent to >500 mg of methylxanthines.
20. Subject has donated or lost ≥450 mL of blood within the previous 2 months prior to study drug administration or has donated plasma within 7 days prior to study drug administration.
21. Known hypersensitivity/allergy reaction to moxifloxacin or other fluoroquinolones.
22. Use of prescription medication within 14 days or 5 half-lives (whichever is longer) or over-the-counter products (including natural food supplements) within 7 days prior to admission to Treatment Period 1, unless in the investigator's opinion the medication does not interfere with the pharmacokinetics of study drug or compromise subject safety. Exceptions include topical products without systemic absorption, hormonal contraceptives, hormone replacement therapy, and acetaminophen (≤2 g/day).
23. Any allergy, intolerance, restriction or special diet that, in the opinion of the investigator, could contraindicate the subject's participation in this study.
24. History of unexplained loss of consciousness, unexplained syncope, unexplained irregular heartbeats or palpitations or near drowning with hospital admission.
25. Subjects who received any investigational drug 30 days or 5 half-lives (whichever is longer) prior to first study drug administration.
26. Use of other forms of nicotine (e-cigarettes, smokeless tobacco) or are planning to use these products during study.
27. Known hypersensitivity/allergy reaction to varenicline, cytisinicline or other cytisinicline-derivatives.
28. Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test, prior to admission to each study period.
29. Any reason which, in the opinion of the investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Predicted Placebo-Adjusted Change From Baseline in the Corrected QT Interval using Fridericia's Formula (QTcF) Interval (ΔΔQTcF) | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.

SECONDARY OUTCOMES:
Placebo-Adjusted Change From Baseline Over Time in Corrected QT Interval (QTc; Corrected for Heart Rate Based on the ΔΔQTcF) | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Placebo-Adjusted Change From Baseline Over Time in Heart Rate (HR) | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Placebo-Adjusted Change From Baseline Over Time in PR Interval of the Electrocardiogram (PR) | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Placebo-Adjusted Change From Baseline Over Time in QRS Interval of the Electrocardiogram (QRS) Duration | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Predicted Placebo-Adjusted Change From Baseline in HR (ΔΔHR) | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Predicted Placebo-Adjusted Change From Baseline in PR (ΔΔPR) | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Predicted Placebo-Adjusted Change From Baseline in QRS Duration (ΔΔQRS) | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Percentage of Participants With New Onset (Post-Baseline) Findings on ECG Morphology | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Uncorrected Change From Baseline Over Time in QT Interval of the Electrocardiogram (QT) | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Uncorrected Change From Baseline Over Time in PR | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Uncorrected Change From Baseline Over Time in QRS | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Uncorrected Change From Baseline Over Time in HR | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.
Percentage of Participants Meeting Outlier Criteria Based on Uncorrected QT, PR, QRS, and HR Values | Day -1 (first treatment period only) and on Day 1 (the day of dosing during each treatment period) from approximately 1 hour pre-dose on Day 1 through approximately 24 hours post dose on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fonseca, MD, Principal Investigator — Blueclinical, Ltd.
Locations (1):
- BlueClinical Phase I, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No